CLINICAL TRIAL: NCT07104760
Title: Longitudinal Evaluation of Regenerative Treatment of Peri-implantitis Assited by Er,Cr:YSGG Laser: up to 10 Years Follow-up
Acronym: Laser
Status: Active, not recruiting | Type: Observational
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Jamil awad shibli, Head, University of Guarulhos
Other Study IDs: Guarulhos University; 2008/07154-5 (Other Grant/Funding Number: FAPESP); #001 (Other Grant/Funding Number: CAPES); 311368/2019-0 (Other Grant/Funding Number: CNPq); 314479/2023-6 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis; Peri-Implantitis and Systemic Inflammation
Keywords: peri-implantitis; surgical treatment
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laser + ATB: Laser-ATB
- LAser_LPR

SUMMARY:
Peri-implantitis is a pathological condition characterized by the inflammation of peri-implant connective tissues and progressive alveolar bone loss. There is a global concern about the increasing prevalence of this disease, which may affect up to 43% of implants in function. This cohort study will evaluated the long term follow up of a randomized, controlled, double-blind placebo study that evaluated the regenerative treatment of peri-implant diseases with surgical debridement and Er,Cr:YSGG AG laser associated with systemic antibiotics. A total of 80 subjects with peri-implantitis (PD>5mm, BoP and/or sup, bone loss >3mm) will be treated reavluated after 10years follow-up. Clinical, radiographic, and microbiological parameters will be recorded at baseline and 120 months follow-up. The primary outcome variable of this trial was be the difference between groups for the change in clinical attachment level from baseline to 6 months. We did consider composite outcomes, although not as the primary outcome. We also aim to evaluate the number and percentage of patients (and implants) reaching the following clinical endpoint for treatment: Probing depth < 5mm, absence of bleeding on probing and no further bone loss (Heitz-Mayfield and Mombelli, 2014). The secondary variables will be the differences between groups in PI, GI, BOP, SUP and PD and microbial profile.

DETAILED DESCRIPTION:
Research design and Methods This double-blinded, two-armed and placebo-controlled study will be conducted at Guarulhos University (UNG; Guarulhos/São Paulo, Brazil). This protocol was elaborated according to the Standard Protocol Items: Recommendations for Interventional Studies (SPIRIT) guidelines (Chan et al. 2013). This trial will be conducted according to the principles of the Declaration of Helsinki for studies in humans. The protocol will be approved by the Institutional Review Board of UNG. All eligible volunteers will be informed about the nature, potential risks and benefits of their participation in this study and will sign a term of free and informed consent.

Subject population and inclusion/exclusion criteria Systemically healthy volunteers with untreated peri-implantitis will be selected from the Oral Implantology Clinic - UNG. Subjects will be selected according to the following inclusion criteria: males and females from 18-70 years old, in general good health, with at least one dental implant in function for at least one year with untreated peri-implantitis defined as: presence of bleeding and/or suppuration on gentle probing, probing depths (PD) ≥ 6 mm, and bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant (Berglundh et al. 2018). The exclusion criteria will be as follows: subjects with ≥ 6 sites with PD ≥5 mm or individuals that received periodontal treatment within three months prior to entering the study, inability to perform proper supramucosal and supragingival plaque control (e.g., due to improper restoration design or lack of skills), poorly adapted implant-supported restoration, diabetes, pregnancy, nursing, history of allergies to MTZ and AMX, or any other ingredient of oral care products, alcohol or drug abuse, any systemic diseases that could affect post-operative healing or that required antibiotic premedication for routine dental therapy, long-term use of mouthrinses, anti-inflammatory medications, or any other drug that could interfere with the study outcomes within three months prior to entering the study and use of antibiotics within six months prior to entering the study.

Interventions At baseline, all volunteers will fill out a structured questionnaire comprised of information about demographic, oral and general health data. Subsequently, they will be submitted to a complete periodontal clinical assessment and collection of submucosal biofilm. In addition, oral hygiene instructions (OHI), full-mouth supramucosal plaque removal, and prophylaxis will be provided. Subgingival scaling will be administered to all sites exhibiting PD ≥4 mm. Partial and total fixed prosthesis on implants will be removed before treatment. Subjects will be given a soft bristle adult toothbrush, dental floss, and interdental toothbrushes, according to their individual needs.

Subsequently, each volunteer will be randomly allocated to one of the following therapeutic groups:

(i) Control: anti-infectious surgical treatment plus placebo. (ii) Test: anti-infectious surgical treatment plus systemic MTZ (400 mg) and AMX (500 mg).

All medications and placebos will be given thrice a day (TID) for 14 days, starting immediately after anti-infectious surgical treatment. Antibiotics and placebos will be specially prepared for this study by the same pharmacy. All tablets will have the same color and size and will be stored in properly coded opaque plastic bottles containing 22 units. Volunteers, personnel (researchers responsible for the treatment) and the examiners will be blind to the intervention. Volunteers will use 21 tablets in the first week and 21 in the second week. Volunteers will not be informed about the total number of tablets in each bottle (22 capsules). They will return the bottles after the first week of treatment and will receive new ones containing the same amount of medication for the second week. Thus, it will be possible to count the number of capsules ingested and the residual capsules (22nd) left in the bottle, in order to monitor compliance. In addition, they will be also monitored every 2 days via telephone. At the end of the medication period (14th day), volunteers will answer a questionnaire about any self-perceived side effects.

The anti-infectious surgical treatment will be performed as follows: after local anesthesia (2% lidocaine with1:100,000 epinephrine), intrasulcular incisions will be performed to create a horizontal flap extending beyond the adjacent teeth and/or implants. Buccal and lingual full-thickness flaps will be dissected, and granulation tissue will be removed to expose the implant threads and bone defect. To remove biofilm and calculus, the implant surface will be scaled and decontaminated with Er:YAG laser. The flap will be repositioned in its original position and stabilized with interrupted sutures, which will be removed after 10 days. Analgesics will be prescribed for all subjects, and they will be instructed to rinse with a 0.12% chlorhexidine mouthwash twice a day for 7 days. The patients will be provided with mouthwashes. All volunteers will receive periodontal maintenance every 2 months post-treatment until the end of the study, including OHI and prophylaxis with ultrasonic scaler and curettes.

Clinical examination One calibrated examiner will perform all clinical examinations. The following parameters will be recorded at six sites per implant and teeth excluding third molars, using a North Carolina periodontal probe (Hu-Friedy, Chicago, IL, USA): Plaque Index (PI) (Quigley & Hein, 1962; Turesky et al., 1970): The plaque will be disclosed using a disclosing solution and recorded as follows: score 0 = absence of plaque; score 1 = separate flecks of plaque on the cervical margin; score 2 = a thin, continuous band of plaque [up to 1 mm] at the cervical margin of the tooth; score 3 = a band of plaque wider than 1 mm, but covering less than 1/3 of the tooth crown; score 4 = plaque covering at least 1/3, but less than 2/3 of the crown of the tooth; score 5 = plaque covering 2/3 or more of the crown of the tooth). Gingival Index (GI) (Loe & Silness, 1963): score 0 = absence of inflammation; score 1 = mild inflammation - change in color and little change in texture; score 2 = moderate inflammation - moderate glazing, redness, edema, and hypertrophy; score 3 = severe inflammation- marked redness and hypertrophy. Tendency to present spontaneous bleeding, presence or absence of bleeding on probing (BOP) and suppuration (SUP), PD (mm), and relative clinical attachment (CA) (distance in mm from the cement-enamel junction/implant shoulder to the most apical portion of the sulcus or periodontal/peri-implant pocket). Implant-supported restorations (screw-retained or cemented) will be removed to allow accurate clinical measurements. A temporary resin restoration will replace cemented implant-supported restoration until the end of the study. The clinical monitoring will be performed at baseline and at time intervals of 3 and 6 months.

Laser Parameters An Er:YAG laser (Lite Touch, Light Instruments, Israel) will be used, with an irradiation energy of 20 mJ, frequency of 20 Hz, output power of 0.4 W, and an energy density of 2.76 J/cm2. An 8 mm long sapphire tip will be used in the respective handpiece and not in contact with the titanium surface, with concomitant water spray irrigation, under air 6 and water spray 6, the irradiation angle will be 90 degrees, at a focal distance of 2 mm, with spot size diameter of 1.3 mm.

Calibration The examiner will be trained and calibrated prior to and during the trial, in order to achieve maximum reproducibility in the measurements. The methodology to be used for the intra-examiner calibration will be that recommended by Araujo et al. (2003), in which the standard error of measurement for continuous periodontal clinical parameters (PD and CAL) is evaluated. For the other clinical variables, the average level of agreement between the examiners will be determined and considered satisfactory when the value is higher than 90% (Kappa test).

Sample size calculation The ideal sample size to assure adequate power for this RCT was calculated considering differences of at least 0.5 mm in CA level (to the mean of 6 sites evaluated in the treated implants) between groups and assuming a standard deviation of 0.8 mm (Stewart et al. 2018, de Mendonça et al. 2009). Based on these calculations, it was defined that 41 subjects per group will be necessary to provide an 80% power with an α of 0.05. Considering an attrition of about 15%, it has been established that at least 47 subjects must be included in each treatment group.

Randomization and allocation concealment An investigator not involved in the inclusion and treatment of the patients will assign the study participants to one of the two treatment groups by means of a computer-generated random sequence (Random Allocation Software, http://random-allocation-software.soft). Randomization will stratify patients according to center with the use of permuted blocks of 3, 6 and 9. In order to assure allocation concealment, the study coordinator will organize the bottles with the tablets in opaque plastic bags labeled with the respective volunteer's number.

ELIGIBILITY:
Inclusion Criteria:

* subjects with peri-implantitis presence of bleeding and/or suppuration on gentle probing, probing depths (PD) ≥ 6 mm, and bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant (Berglundh et al. 2018); treated by one of the treatment groups

Exclusion Criteria:

* failed implants, subjects with pregnancy or oncological problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically healthy volunteers with treated peri-implantitis will be selected from the Oral Implantology Clinic - UNG.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | 120 months
  CAL mm
CAL | 10 years
  gain of 1mm CAL

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Shibli, PhD, Principal Investigator — University of Guarulhos
Locations (1):
- Guarulhos University, Guarulhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
under consideration after IRB approval